CLINICAL TRIAL: NCT06462183
Title: A Phase 1a/1b, First-in-human, Multicenter Study to Assess the Efficacy and Safety of RGT-61159 for Treatment of Patients With Relapsed/Refractory Adenoid Cystic Carcinoma (ACC) or Colorectal Carcinoma (CRC)
Brief Title: Study of Safety and Efficacy of RGT-61159 in Adults With Relapsed/Refractory Adenoid Cystic Carcinoma (ACC) or Colorectal Carcinoma (CRC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rgenta Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGT61159-01
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Adenoid Cystic Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, ascending dose escalation followed by dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): RGT-61159 in escalating doses
  Interventions: Drug: RGT-61159
- Dose expansion Cohort A (Experimental): Dose optimization; RGT-61159, 2 doses, randomized allocation
  Interventions: Drug: RGT-61159
- Dose expansion Cohort B (Experimental): Simon's 2 stage, RGT-61150 at optimized dose from Part A
  Interventions: Drug: RGT-61159

INTERVENTIONS:
Drug: RGT-61159 — Oral MYB inhibitor

SUMMARY:
Phase 1 study to evaluate safety, tolerability and anti-tumor activity of RGT-61159 in patients with ACC or CRC

DETAILED DESCRIPTION:
This first-in-human, Phase 1, multi-center, open-label, non-randomized study, is designed to evaluate safety, tolerability, and anti-tumor activity of once-daily RGT-61159 in patients with advanced R/R ACC or R/R CRC for whom standard therapy with proven clinical benefit does not exist, is no longer effective, or is not appropriate. RGT-61159 is an oral, small molecule MYB inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ACC or CRC
* Radiographically measurable disease as assessed per RECIST 1.1, with at least 1 site of disease that is measurable and that has not been previously irradiated; or, if the patient has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation
* Patients with locally relapsed/refractory (R/R) advanced or metastatic ACC not amenable to potentially curative surgery or radiotherapy and progression of disease within 12 months at study entry
* Patients with CRC must have locally R/R advanced or metastatic disease not amenable to potentially curative surgery or radiotherapy; must have been previously treated with, or are not considered candidates for, available therapies including fluoropyrimidines-, oxaliplatin-, and irinotecan-based chemotherapies, anti-VEGF agents, and if RAS wild-type, an anti-EGFR therapy.
* Adequate hematologic status, organ function, renal function, liver function and prothrombin time (PT) or INR ≤ 1.5 × ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Resolved acute effects of any prior therapy to baseline

Exclusion Criteria:

* Major surgery or significant traumatic injury within 28 days prior to Cycle 1 Day 1
* Chemotherapy within 14 days prior to Cycle 1 Day 1
* Use of nitrosoureas or mitomycin C within 6 weeks prior to Cycle 1 Day 1
* Radiation therapy within 21 days prior to Cycle 1 Day 1
* Investigational drug use, targeted therapy, or biologic therapy within 28 days or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1
* Ongoing systemic infection requiring treatment with antibiotic, antiviral, or antifungal treatment
* Active known second malignancy
* Clinically significant cardiac disease
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2 unless it's well-controlled HIV (eg, cluster of differentiation 4 [CD4] > 350/mm3 and undetectable viral load)
* Current active liver disease including hepatitis A (hepatitis A [HepA] virus immunoglobulin M [IgM] positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV RNA)
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate absorption
* Uncontrolled diabetes
* Treatment with a long-acting hematopoietic growth factor within 14 days before Cycle 1 Day 1 or a short-acting hematopoietic growth factor within 7 days before Cycle 1 Day 1
* Treatment with high-dose chemotherapy and stem-cell rescue (autologous stem cell transplant) or allogeneic stem cell transplant within 90 days before Cycle 1 Day 1
* Patients with central nervous system (CNS) metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroid throughout this indication for at least 4 weeks before starting treatment in this study
* History of solid organ transplantation
* Coronavirus disease 2019 (COVID-19) vaccination within 14 days prior to first dose of study drug
* Prior treatment with a MYB inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number and type of dose-limiting toxicities (DLTs) in first cycle of administration | 21 days
Number and type of adverse events | Through study completion, estimated as 30 days after last dose of study drug
Recommended Phase 2 Dose (RP2D) | Assessed at the end of Cycle 1 for each subject (each cycle 21 days)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology VA, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (2):
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No